CLINICAL TRIAL: NCT02883504
Title: Validation Study of the Accuracy of E/e' in Estimating Left Ventricular Filling Pressure
Acronym: EUROFILLING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01331-46; 35RC14_3003 (Other: CHU Rennes)
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Doppler Echocardiography
Keywords: E/e' ratio; Doppler echocardiography, filling pressure; Left Ventricular end-Diastolic Pressure

ARMS (1):
- Echocardiography (Experimental)
  Interventions: Procedure: Echo-Doppler examination and left heart catheterization

INTERVENTIONS:
Procedure: Echo-Doppler examination and left heart catheterization

SUMMARY:
The non-invasive estimation of left ventricular end diastolic pressure (LVeDP) is a main goal for performing an echocardiography in the routine clinical practice. Conflicting evidence exists about mitral E/e' ratio reliability for predicting high LVeDP

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient performing an echocardiography in the routine clinical practice
* Informed consent given

Exclusion Criteria:

* Severe valve disease, valvular prostheses, calcification of the mitral valve, the history of myocardial infarction, atrial fibrillation, severe arrhythmias not allowing the Doppler analysis, pacemaker and any image by inadequate Doppler ultrasound
* Major person under legal protection (backup justice, trusteeship, guardianship), person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Invasive evaluation of left ventricular end diastolic pressure | D0
  Left heart catheterization

SECONDARY OUTCOMES:
Non-invasive evaluation of left ventricular end diastolic pressure | D0
  Echo-Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, Md, PhD, Study Director — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France